CLINICAL TRIAL: NCT01438255
Title: Observational Study on Efficacy of Alvesco(Ciclesonide) in Asthma Children and Adolescent in Real Practice
Status: Completed | Type: Observational
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALVESCO-OS01
Record Dates: First submitted 2011-09-08; First posted 2011-09-22 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Alvesco

SUMMARY:
This is a prospective, non-comparative, open, observational study.

ELIGIBILITY:
Inclusion Criteria:

* Children who is prescribed with ciclesonide for asthma

Exclusion Criteria:

* Subjects with contraindications to ciclesonide use
* Subjects with clinically relevant concomitant disease that could compromise the patient's safety should not be included in this study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: outpatients
Sampling Method: Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Asthma control day | 12weeks

SECONDARY OUTCOMES:
Morning peak expiratory flow | 12weeks
asthma exacerbation | 12weeks
The number of Reliever use | 12weeks
Asthma symptom score | 12weeks
Number of Participants with Adverse Events | 12weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Handok Pharmaceuticals, Seoul, Seoul, South Korea